CLINICAL TRIAL: NCT00853242
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study Using Genz-644470 and Sevelamer Carbonate in Hyperphosphatemic Chronic Kidney Disease Patients on Hemodialysis
Brief Title: Randomized Study Comparing Genz-644470, Placebo, and Sevelamer Carbonate in Chronic Kidney Disease Patients on Hemodialysis
Acronym: LEAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APB00108
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Kidney Failure, Chronic
Keywords: Chronic Kidney Disease; Phosphate Binder; Phosphate; Hyperphosphatemia
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator): Placebo matched to Genz-644470 tablet orally three times a day (TID) with meals for 3 weeks.
  Interventions: Drug: Placebo
- Genz-644470 2.4 Grams Per Day (g/day) (Experimental): Genz-644470 2.4 g/day tablets dosed orally TID with meals for 3 weeks.
  Interventions: Drug: Genz-644470
- Genz-644470 4.8 g/day (Experimental): Genz-644470 4.8 g/day tablets dosed orally TID with meals for 3 weeks.
  Interventions: Drug: Genz-644470
- Genz-644470 7.2 g/day (Experimental): Genz-644470 7.2 g/day tablets dosed orally TID with meals for 3 weeks.
  Interventions: Drug: Genz-644470
- Sevelamer Carbonate 2.4 g/day (Active Comparator): Sevelamer Carbonate 2.4 g/day tablets dosed orally TID with meals for 3 weeks.
  Interventions: Drug: Sevelamer carbonate
- Sevelamer Carbonate 4.8 g/day (Active Comparator): Sevelamer Carbonate 4.8 g/day tablets dosed orally TID with meals for 3 weeks.
  Interventions: Drug: Sevelamer carbonate
- Sevelamer Carbonate 7.2 g/day (Active Comparator): Sevelamer Carbonate 7.2 g/day tablets dosed orally TID with meals for 3 weeks.
  Interventions: Drug: Sevelamer carbonate

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Genz-644470
  Arms: Genz-644470 2.4 Grams Per Day (g/day); Genz-644470 4.8 g/day; Genz-644470 7.2 g/day
Drug: Sevelamer carbonate
  Other Names: Renvela®
  Arms: Sevelamer Carbonate 2.4 g/day; Sevelamer Carbonate 4.8 g/day; Sevelamer Carbonate 7.2 g/day

SUMMARY:
The purpose of this clinical study is to compare the effects of Genz-644470 with the effects of placebo and sevelamer carbonate (Renvela®) on the reduction of serum phosphorus in hyperphosphatemic chronic kidney disease participants on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Serum phosphate level greater than (>) 5.5 milligram per deciliter (mg/dL) (1.78 millimole per liter [mmol/L]) after discontinuation of current phosphate binder therapy
* Men or women 18 years or older

Exclusion Criteria:

* Have active dysphagia or swallowing disorder or a predisposition to or current bowel obstruction, ileus, or severe gastrointestinal motility disorders including severe constipation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (53):
- United States (52):
  - Alexander City, Alabama
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Bakersfield, California
  - Los Angeles, California
  - Paramount, California
  - Pembroke Pines, California
  - Porterville, California
  - Riverside, California
  - San Dimas, California
  - Whittier, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Hudson, Florida
  - Ocala, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Marietta, Georgia
  - Gurnee, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Bethesda, Maryland
  - Pontiac, Michigan
  - Southfield, Michigan
  - Brookhaven, Mississippi
  - Gulfport, Mississippi
  - St Louis, Missouri
  - Kearney, Nebraska
  - Las Vegas, Nevada
  - Bellmore, New York
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Port Washington, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Cincinnati, Ohio
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Lewistown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Columbia, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Alexandria, Virginia
  - Glendale, Wisconsin
  - Milwaukee, Wisconsin
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 64 centers in the United States between 11 February 2009 and 20 August 2009.
Pre-assignment Details: A total of 670 participants were screened of which 321 were screen failure and 349 participants were randomized. After screening, participants entered a two-week phosphate binder washout period prior to randomization.
Period: Overall Study
Arm/Group | Placebo | Genz-644470 2.4 Grams Per Day (g/Day) | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day | Sevelamer Carbonate 2.4 g/Day | Sevelamer Carbonate 4.8 g/Day | Sevelamer Carbonate 7.2 g/Day
Started | 50 | 50 | 49 | 50 | 50 | 51 | 49
Treated | 50 | 49 | 48 | 50 | 50 | 51 | 48
Completed | 47 | 47 | 46 | 46 | 46 | 49 | 44
Not Completed | 3 | 3 | 3 | 4 | 4 | 2 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 3 | 1 | 1
Not completed — Noncompliant | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 4 | 0 | 0 | 2
Not completed — Other | 2 | 0 | 2 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set included all randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Placebo matched to Genz-644470 tablet orally TID with meals for 3 weeks.
- Genz-644470 2.4 g/Day: Genz-644470 2.4 g/day tablets dosed orally TID with meals for 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Genz-644470 2.4 g/Day | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day | Sevelamer Carbonate 2.4 g/Day | Sevelamer Carbonate 4.8 g/Day | Sevelamer Carbonate 7.2 g/Day | Total
Number analyzed (Participants) | 50 | 49 | 48 | 50 | 50 | 51 | 48 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (13.6) | 58.3 (12.0) | 54.7 (11.3) | 56.7 (13.3) | 54.6 (13.4) | 56.6 (11.9) | 53.6 (13.1) | 56.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 23 | 19 | 22 | 21 | 15 | 144
  Male | 30 | 25 | 25 | 31 | 28 | 30 | 33 | 202
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 1 | 1 | 2 | 0 | 2 | 8
  Black or African American | 21 | 20 | 25 | 25 | 23 | 25 | 22 | 161
  White | 29 | 27 | 22 | 22 | 25 | 25 | 23 | 173
  Other | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 4
Serum Phosphorus Level [Number; unit: participants]
  less than (<) 7.0 milligram per deciliter (mg/dL) | 22 | 22 | 21 | 21 | 22 | 20 | 17 | 145
  Greater Than or Equal to (>=) 7.0 mg/dL | 28 | 27 | 27 | 29 | 28 | 31 | 31 | 201

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Phosphorus at Day 22 (Genz-644470 vs Placebo)
Time Frame: Baseline, Day 22
Population: Full Analysis Set (FAS) included all participants who received at least one dose of study drug and had baseline and at least one post-baseline phosphorus measure less than or equal to (<=) 3 days after date of last study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Genz-644470 2.4 g/Day | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day
Number analyzed (Participants) | 50 | 48 | 47 | 46
mg/dL | -0.0 (1.3) | -0.6 (1.5) | -1.2 (1.6) | -1.8 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Genz-644470 2.4 g/Day; Analysis was performed using Wilcoxon rank sum tests; Test type: Superiority or Other; p = 0.0249, Wilcoxon Rank Sum Tests
Statistical Analysis 2: Comparison: Placebo vs Genz-644470 4.8 g/Day; Analysis was performed using Wilcoxon rank sum tests; Test type: Superiority or Other; p = 0.0001, Wilcoxon Rank Sum Tests
Statistical Analysis 3: Comparison: Placebo vs Genz-644470 7.2 g/Day; Analysis was performed using Wilcoxon rank sum tests; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Tests

2. Secondary Outcome: Change From Baseline in Serum Phosphorus at Day 22 (Genz-644470 vs Sevelamer Carbonate)
Time Frame: Baseline, Day 22
Population: FAS included all participants who received at least one dose of study drug and had baseline and at least one post-baseline phosphorus measure <= 3 days after date of last study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Genz-644470 2.4 g/Day | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day | Sevelamer Carbonate 2.4 g/Day | Sevelamer Carbonate 4.8 g/Day | Sevelamer Carbonate 7.2 g/Day
Number analyzed (Participants) | 48 | 47 | 46 | 49 | 48 | 47
mg/dL | -0.6 (1.5) | -1.2 (1.6) | -1.8 (1.9) | -0.9 (1.7) | -1.3 (1.9) | -2.0 (1.4)
Statistical Analysis 1: Comparison: Genz-644470 2.4 g/Day vs Sevelamer Carbonate 2.4 g/Day; Analysis was performed using Wilcoxon rank sum tests; Test type: Superiority or Other; p = 0.2647, Wilcoxon Rank Sum Tests
Statistical Analysis 2: Comparison: Genz-644470 4.8 g/Day vs Sevelamer Carbonate 4.8 g/Day; Analysis was performed using Wilcoxon rank sum tests; Test type: Superiority or Other; p = 0.7944, Wilcoxon Rank Sum Tests
Statistical Analysis 3: Comparison: Genz-644470 7.2 g/Day vs Sevelamer Carbonate 7.2 g/Day; Analysis was performed using Wilcoxon rank sum tests; Test type: Superiority or Other; p = 0.3724, Wilcoxon Rank Sum Tests

3. Secondary Outcome: Change From Baseline in Serum Calcium (Albumin-adjusted)-Phosphorus Product at Week 22
Time Frame: Baseline, Day 22
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg^2/dL^2
Arm/Group | Placebo | Genz-644470 2.4 g/Day | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day | Sevelamer Carbonate 2.4 g/Day | Sevelamer Carbonate 4.8 g/Day | Sevelamer Carbonate 7.2 g/Day
Number analyzed (Participants) | 50 | 48 | 47 | 46 | 49 | 48 | 47
mg^2/dL^2 | -0.1 (12.7) | -4.5 (12.3) | -9.2 (14.7) | -16.1 (16.1) | -8.3 (17.4) | -10.3 (17.5) | -17.5 (13.4)

4. Secondary Outcome: Change From Baseline in Total Cholesterol at Day 22
Time Frame: Baseline, Day 22
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Genz-644470 2.4 g/Day | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day | Sevelamer Carbonate 2.4 g/Day | Sevelamer Carbonate 4.8 g/Day | Sevelamer Carbonate 7.2 g/Day
Number analyzed (Participants) | 50 | 48 | 47 | 46 | 49 | 48 | 47
mg/dL | -3.8 (20.9) | -13.5 (20.7) | -11.2 (19.7) | -17.8 (22.8) | -2.9 (17.1) | -15.8 (16.3) | -18.1 (27.8)

5. Secondary Outcome: Change From Baseline in Low Density Lipoprotein (LDL) Cholesterol at Day 22
Time Frame: Baseline, Day 22
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Genz-644470 2.4 g/Day | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day | Sevelamer Carbonate 2.4 g/Day | Sevelamer Carbonate 4.8 g/Day | Sevelamer Carbonate 7.2 g/Day
Number analyzed (Participants) | 50 | 48 | 47 | 46 | 49 | 48 | 47
mg/dL | -1.3 (17.4) | -15.4 (19.8) | -13.2 (18.6) | -21.9 (23.5) | -7.5 (13.0) | -17.7 (14.8) | -22.6 (24.5)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Day 22) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the first dose of study drug up to 30 days after last dose of study drug). The Safety Set included all randomized participants who were treated with at least one dose of study drug.
Arm/Group | Placebo | Genz-644470 2.4 g/Day | Genz-644470 4.8 g/Day | Genz-644470 7.2 g/Day | Sevelamer Carbonate 2.4 g/Day | Sevelamer Carbonate 4.8 g/Day | Sevelamer Carbonate 7.2 g/Day
Serious Adverse Events (participants affected / at risk) | 4/50 | 2/49 | 6/48 | 6/50 | 8/50 | 5/51 | 5/48
Other Adverse Events (participants affected / at risk) | 17/50 | 17/49 | 17/48 | 25/50 | 22/50 | 25/51 | 22/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | Genz-644470 2.4 g/Day (N=49) | Genz-644470 4.8 g/Day (N=48) | Genz-644470 7.2 g/Day (N=50) | Sevelamer Carbonate 2.4 g/Day (N=50) | Sevelamer Carbonate 4.8 g/Day (N=51) | Sevelamer Carbonate 7.2 g/Day (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arteriovenous graft site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Catheter bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal transplant (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | Genz-644470 2.4 g/Day (N=49) | Genz-644470 4.8 g/Day (N=48) | Genz-644470 7.2 g/Day (N=50) | Sevelamer Carbonate 2.4 g/Day (N=50) | Sevelamer Carbonate 4.8 g/Day (N=51) | Sevelamer Carbonate 7.2 g/Day (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 1 | 4 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 3 | 2 | 3 | 7
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 2 | 3
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0
Catheter related complication (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 4 | 1 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.